CLINICAL TRIAL: NCT01793519
Title: Stopping Tumor Necrosis Factor-Alpha Inhibitors in Rheumatoid Arthritis (STARA) Clinical Trial
Brief Title: Stopping TNF Alpha Inhibitors in Rheumatoid Arthritis
Acronym: STARA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); University of Maryland, Baltimore (Other); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); Medstar Health Research Institute (Other); Patient-Centered Outcomes Research Institute (Other); Arthritis and Pain Associates of PG County (Unknown); Arthritis & Rheumatism Associates, P.C. (Other); Rheumatology Associates of Baltimore, L.L.C. (Unknown); The Arthritis Clinic of Northern Virginia, P.C. (Unknown); Arthritis and Rheumatic Disease Associates, P.C. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER-1402-10522; 13-AR-0056 (Other: Internal NIAMS assigned number); CER-1402-10522 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Autoimmune Diseases; Anti-TNF
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases | interventions — Etanercept; Infliximab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anti-tumor necrosis factor agent (Active Comparator): Anti-TNF agent - etanercept, infliximab, adalimumab - administered parentally at standard dosage and frequencies
  Interventions: Drug: Etanercept; Drug: Infliximab; Drug: Adalimumab
- Placebo (Placebo Comparator): Administered appropriately to active comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etanercept — Subcutaneous
  Other Names: Enbrel
  Arms: Anti-tumor necrosis factor agent
Drug: Infliximab — Infusion
  Other Names: Remicade
  Arms: Anti-tumor necrosis factor agent
Drug: Adalimumab — Subcutaneous
  Other Names: Humira
  Arms: Anti-tumor necrosis factor agent
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
Background:

* Rheumatoid arthritis (RA) is often treated with drugs known as tumor necrosis factor (TNF) inhibitors, that can help decrease joint pain and swelling and can even result in RA remission. However, TNF inhibitors may increase risk of serious infections or some types of cancer.
* It is not clear if people whose RA has been in remission for a long time need to stay on the TNF inhibitor to remain in remission. If they can stop taking the TNF inhibitor without having their symptoms come back, they will be spared the side effects of these medicines. Some studies have shown that people can stay in remission after stopping a TNF inhibitor, but other studies have not confirmed it. Researchers want to see if people with RA in remission on a TNF inhibitor can stay in remission without this medicine. Also there may be a clinical, imaging (MRI, ultrasound), laboratory profile that will help to determine which patients remain in remission after stopping these drugs.

Objectives:

* To see whether RA remission can continue after discontinuing use of a TNF inhibitor.
* To determine if clinical, imaging and immunological measurements can predict which participants will flare and which will remain in remission after discontinuing TNF inhibitor.

Eligibility:

-Individuals at least 18 years of age who have RA that is being controlled with TNF inhibitors. We plan to randomize 291 patients.

Design:

* The study has seven visits over about 2 years. Six visits occur in the first year of the study, about 12 weeks apart. The final study visit is 1 year after the end of the treatment phase.
* At the first visit, participants will be screened with a physical exam and medical history. They will complete a questionnaire about their RA symptoms. A blood sample will be collected. They will continue to take their RA medicines during this time.
* The second visit will repeat tests from the first visit. These tests will confirm that the RA is in remission. Imaging studies will be performed on the hands, wrists, feet, and their connected joints. After this visit, participants will stop taking their TNF inhibitors and will start to have injections of a study drug. This drug will be either the participant's original TNF inhibitor or a placebo.
* There will be follow-up visits at weeks 12, 24, and 36. Participants will have a medical history and joint exam. They will also provide blood samples and answer questions about their RA symptoms.
* At the sixth visit (week 48), participants will repeat the tests and imaging studies from the second visit. They will stop taking the study injections.
* Continued RA treatment after this visit will be decided by the participant and his or her rheumatologist. Participants may take any recommended medicine, including the TNF inhibitor they had been taking before the study. They will also receive a questionnaire to complete at home and mail back before the final study visit.
* At the final visit (week 100), participants will repeat the tests and imaging studies from the second and sixth visits.

DETAILED DESCRIPTION:
Remission of rheumatoid arthritis (RA) is an achievable goal with currently available medications, including the anti-tumor necrosis factor (anti-TNF) agents. However, it is uncertain if patients with RA in clinical remission while treated with anti-TNF agents and background disease-modifying antirheumatic drugs (DMARD) would remain in remission if anti-TNF therapy was stopped. If remission can be sustained off anti-TNF agents, then patients may be spared the potential toxicity and costs of these medications.

The Stopping Anti-Tumor Necrosis Factor Agents in Rheumatoid Arthritis (STARA) study is a multicenter, randomized, double-blind, placebo-controlled noninferiority trial that will test differences in time to relapse between patients with RA in remission who discontinue anti-TNF agents and patients with RA in remission who continue anti-TNF agents. The secondary objectives of the study are: 1) to determine if discontinuation of anti-TNF agents results in a difference in progression of joint damage on radiographs; 2) to determine if discontinuation of anti-TNF agents results in a difference in physical function, and 3) to identify predictors of relapse.

Eligible subjects will have RA in remission for at least six months while taking etanercept, infliximab, or adalimumab. An eight-week run-in period prior to randomization will be used to confirm remission. Subjects will then be randomized in a 2:1 ratio to receive one of two blinded treatments: 1) matching placebo or 2) their currently used anti-TNF agent, respectively. All subjects will maintain their current background DMARD. Clinical assessments will be performed every 12 weeks. The primary outcome is 48-week relapse-free status. Secondary outcomes include change from baseline radiographic joint damage score at 48 weeks and 100 weeks, and change from baseline physical function score at 48 weeks. Subjects who relapse before week 48 will discontinue study medication and receive treatment through their rheumatologist. Blinded treated will end at week 48 and subjects will be followed for 52 additional weeks. This study will provide important new information on the best treatment approach for patients with RA in remission.

ELIGIBILITY:
* Study personnel will evaluate participant eligibility using a checklist of inclusion and exclusion criteria as outlined below. Clinical information will be obtained from subjects by interview and from the medical record.

At the screening visit, potential participants will be included if:

* Age greater than or equal to 18 years
* Have RA, as defined by the 1987 revised American College of Rheumatology criteria
* In sustained clinical remission for the last 6 months while receiving treatment with either etanercept, infliximab, or adalimumab, and greater than or equal to 1 DMARD (methotrexate, hydroxychloroquine, sulfasalazine, leflunomide, minocycline, cyclosporine, azathioprine, gold, penicillamine). DAS28 should be less than 2.6 on each visit over the preceding 6 months, with at least one visit 2-4 months before enrollment. If there is no visit 6 months before enrollment, the nearest visit in the 6-12 month period before enrollment should be considered and have a DAS28 less than 2.6.

Potential participants will be excluded if:

* Had dose increase of anti-TNF agent or DMARD in the last 6 months
* Had change of anti-TNF agent or DMARD in the last 6 months
* Treated currently with golimumab or certolizumab
* Treated with greater than 10 mg of prednisone (or equivalent) daily in the last 6 months
* Treated with greater than 5 mg of prednisone (or equivalent) daily in the last 3 months
* Treated with intramuscular or intravenous corticosteroids in the last 6 months for RA activity
* Treated with anakinra, abatacept, or tocilizumab in the last 6 months
* Treated with rituximab in the last 12 months
* Treated with an investigational RA drug in the last 6 months
* Pregnant (or anticipate pregnancy during the study period) or lactating women
* Absence of documentation in the medical record of clinical remission for the last 6 months
* Unwilling to discontinue anti-TNF agent
* Absence of documentation of negative tuberculin skin test, negative QuantiFERON-TB Gold test, or treatment for latent tuberculosis prior to starting treatment with the anti-TNF agent
* Treatment of solid malignancy or non-melanoma skin cancer within the past 5 years, or any history of melanoma or hematologic or lymphoproliferative malignancy
* Absence of documentation of age-appropriate cancer screening at the time of randomization
* Absence of documentation of negative hepatitis B serologies, absence of completion of treatment for chronic hepatitis B, or absence of suppressive antiviral treatment
* Unable to provide informed consent
* Anticipate not being available or able to comply with the schedule of study visits

Study entry is not limited by gender or ethnicity. Children are excluded because inflammatory polyarthritis developing before age 16 is considered juvenile idiopathic arthritis and not RA. Patients who developed RA while age 17 would be eligible, but given the time needed to achieve remission, these patients would in most cases be 18 or older by the time they would meet other criteria for study entry.

Participants will largely be recruited from the practices of study investigators. To identify potential subjects, investigators may search rosters of patients in their practice for patients who meet the inclusion criteria. The number of patients screened and reasons for exclusion will be tabulated at each site. Subjects may also be recruited by physician referral. Information about the study will be mailed to local rheumatologists and posted on the NIAMS website. We do not anticipate self-referral of subjects but eligible self-referred subjects will not be excluded.

During the course of the study, enrollment of subjects treated with a particular anti-TNF agent may be suspended or terminated to permit adequate representation of patients treated with each of the 3 anti-TNF medications, due to problems procuring medication, or due to other unforeseen issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2013-01; Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Remission by Disease Activity Score - 28 over 48 weeks | 48 weeks

SECONDARY OUTCOMES:
Change in Health Assessment Questionnaire Disability Index over 48 weeks | 48 weeks
Change in Sharp-van der Heijde radiographic score over 48 weeks | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Ward, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS); Florina Constantinescu, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choy EH, Panayi GS. Cytokine pathways and joint inflammation in rheumatoid arthritis. N Engl J Med. 2001 Mar 22;344(12):907-16. doi: 10.1056/NEJM200103223441207. No abstract available. PMID 11259725
- [Background] Lawrence RC, Helmick CG, Arnett FC, Deyo RA, Felson DT, Giannini EH, Heyse SP, Hirsch R, Hochberg MC, Hunder GG, Liang MH, Pillemer SR, Steen VD, Wolfe F. Estimates of the prevalence of arthritis and selected musculoskeletal disorders in the United States. Arthritis Rheum. 1998 May;41(5):778-99. doi: 10.1002/1529-0131(199805)41:53.0.CO;2-V. PMID 9588729
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Derived] Ward MM, Weinstein A, Alejandro-Silva P, Matsumoto AK, Konatalapalli R, Stahl N, Kerr GS, Mikdashi J, Kempf P, Shah NR, Danielides S, Ghafouri M, Olenginski TP, Fike A, Balyozova-Dinkov D, Thiele R, Yao L, Paul S, Constantinescu F. Discontinuation versus continuation of maintenance treatment with tumor necrosis factor inhibitors in patients with rheumatoid arthritis with low disease activity or remission: A randomized double-blind placebo-controlled trial. Semin Arthritis Rheum. 2025 Dec;75:152831. doi: 10.1016/j.semarthrit.2025.152831. Epub 2025 Sep 17. PMID 41045868
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-AR-0056.html